CLINICAL TRIAL: NCT06083610
Title: Investigation of MicroRNA-1 (miRNA-1) and MicroRNA-133a (miRNA-133a) Levels After Acute Neuromuscular Exercise in Ultimate Frisbee Athletes
Brief Title: MicroRNA-1 (miRNA-1) and MicroRNA-133a (miRNA-133a) Levels After Acute Exercise in Ultimate Frisbee Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Mehmet Alperen Pekdaş, Research Assistant, Yeditepe University
Other Study IDs: 14
Record Dates: First submitted 2023-09-18; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: To Determine the Levels of miRNA1 and miRNA133a Before and After Exercise
Keywords: microRNA; acute exercise; skeletal muscle; exercise training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: miRNA levels analysis from saliva samples — Each participant will be given two 50-mL Falcon tubes and will be asked to expectorate a small amount (about 1 mL) of saliva before and immediately after the end of exercise. Part of each saliva sample will be mixed with an equal volume of denaturing solution included in the mirVanaTM PARISTM kit from Ambion, Foster City, CA, in order to inactivate ribonucleases. Serum samples will be separated by centrifugation at 4000 rpm from the saliva samples taken into the biochemistry tubes of the participants and controls and will be raised to -80 centigrade degrees until the study day. Micro RNA will be isolated from serum samples on the working day. Determination of microRNA expression levels (micro RNA-1 and micro RNA-133a) will be determined by reverse transcriptase polymerase chain reaction (RT-PCR) (Applied Biosystems 7500 Fast Real-Time PCR).

SUMMARY:
"The goal of this clinical trial is to investigate the levels of microRNA-1 (miRNA-1) and microRNA-133a (miRNA-133a) after acute neuromuscular exercise (NME) in human saliva.

The main questions it aims to answer are:

* How do miRNA-1 and miRNA-133a levels change in response to acute neuromuscular exercise in human saliva?
* Will the chosen training method have an acute effect in ultimate frisbee athletes?

Participants will:

* Undergo acute neuromuscular exercise (NME).
* Provide saliva samples for miRNA analysis.

Researchers will compare:

MiRNA-1 and miRNA-133a levels before and after acute neuromuscular exercise (NME) to determine if exercise induces any significant changes in these microRNA levels."

DETAILED DESCRIPTION:
The genetic material in humans and other living things is DNA, and the information in DNA is transcribed into RNA, and RNA translates this information into protein through translation. More than 98% of RNA cannot be translated into protein this untranslated part is called non-coding RNA. Of the non-coding RNAs, micro-RNAs (miRNAs) are short RNAs of approximately 21-23 nucleotides in length that do not code for proteins and that control gene expression after transcription. miRNAs can partially bind to target messenger RNAs (mRNAs), suppressing protein production or silencing gene expression by splicing target mRNAs. miRNAs enable cell differentiation and development by using the translational repression mechanism. In addition to these roles, miRNAs play a role in many points such as cellular metabolism, repair mechanisms, signaling, cell division, and apoptosis pathways. Studies also identify miRNAs as essential intracellular mediators of processes involved in exercise adaptation, including angiogenesis, inflammation, mitochondrial metabolism, cardiac and skeletal muscle contraction force generation, and tissue hypertrophy. There is evidence that the miRNA may play an important role in regulating the plasticity of the skeletal muscles, such as the hypertrophy of the skeletal muscles, or in regulating the functional properties of the muscle. More than 2000 miRNAs have been identified in humans, and some of them are found and function in the human body in a tissue-specific manner. For example, miRNAs, mostly found in muscle tissue and therefore called myomiRs, are involved in proliferation, muscle cell differentiation, metabolism, and hypertrophy in skeletal and cardiac muscles. The myomiR class includes miR-1, miR-133a, miR-133b, miR-206, miR-208a, miR-208b, miR-486, and miR-499. In the literature, studies examine miRNA levels before and after using various exercise modalities. It has been stated that different miRNAs provide responses such as ventricular compliance, hypertrophy, angiogenesis, and mitochondrial biogenesis after acute or chronic exercise. It has been shown in many studies that these responses, decreased or increased miRNA levels after exercise, are related to the target genes they affect, such as IGF-1, PGC-1α, MAPK, TGF-β, COL1A1, and FOXJ3.

The aim of the study is to investigate the levels of miRNA-1 and miRNA-133a levels after acute neuromuscular exercise (NME) in human saliva.

ELIGIBILITY:
Inclusion Criteria:

* Not suffering from an acute illness
* Not having had an orthopedic injury in the last 12 weeks may prevent them from exercising
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of an acute disease
* Having an orthopedic injury that may prevent exercise in the last 12 weeks
* Regular use of medication and/or dietary supplements
* Presence of a chronic & systemic disease
* Not volunteering to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ultimate Frisbee team athletes of a university
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Determination of miRNA-1 and miRNA-133a levels before and after acute neuromuscular exercise | Approximately 1.5 hours for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Turgay İsbir, Prof. Dr., Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Safdar A, Abadi A, Akhtar M, Hettinga BP, Tarnopolsky MA. miRNA in the regulation of skeletal muscle adaptation to acute endurance exercise in C57Bl/6J male mice. PLoS One. 2009;4(5):e5610. doi: 10.1371/journal.pone.0005610. Epub 2009 May 19. PMID 19440340
- [Result] McCarthy JJ, Esser KA. MicroRNA-1 and microRNA-133a expression are decreased during skeletal muscle hypertrophy. J Appl Physiol (1985). 2007 Jan;102(1):306-13. doi: 10.1152/japplphysiol.00932.2006. Epub 2006 Sep 28. PMID 17008435
- [Result] Ultimo S, Zauli G, Martelli AM, Vitale M, McCubrey JA, Capitani S, Neri LM. Influence of physical exercise on microRNAs in skeletal muscle regeneration, aging and diseases. Oncotarget. 2018 Mar 30;9(24):17220-17237. doi: 10.18632/oncotarget.24991. eCollection 2018 Mar 30. PMID 29682218